CLINICAL TRIAL: NCT05929872
Title: The Efficacy of Strategic Memory Training Coupled With Non-invasive Brain Stimulation Techniques in Healthy Aging Population and Subjective Cognitive Decline Patients: a Randomized-controlled Study
Brief Title: Non-invasive Brain Stimulation and Strategic Memory Training
Acronym: StMe-tDCS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS National Neurological Institute "C. Mondino" Foundation (Other)
Collaborators: University of Pavia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: StMe-tDCS2023
Record Dates: First submitted 2023-06-16; First posted 2023-07-03 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: Cognitive Decline; Healthy Aging
Keywords: Healthy aging; Subjective cognitive decline; Non-pharmacological treatments; Memory training; Transcranial direct current stimulation
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: Prospective, double-blind, randomized controlled study
Who Masked: Participant, Investigator
Masking Description: Double
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): The experimental group receives strategic memory training plus non-invasive brain stimulation (ACTIVE tDCS).
  Interventions: Other: Non-invasive brain stimulation
- Control Group (Sham Comparator): The control group receives strategic memory training plus sham non-invasive brain stimulation (SHAM tDCS).
  Interventions: Other: Sham non-invasive brain stimulation

INTERVENTIONS:
Other: Non-invasive brain stimulation — ACTIVE transcranial direct current stimulation( tDCS)
  Arms: Experimental group
Other: Sham non-invasive brain stimulation — SHAM tDCS
  Arms: Control Group

SUMMARY:
Physiological aging is often associated with memory function decline. Recently, the use of transcranial direct current stimulation (tDCS), a type of non-invasive brain stimulation, has been combined with adaptive working memory training interventions in healthy older adults, providing evidence for a significant improvement in memory functions. To the best of our knowledge, no study addressed the use of strategic memory training coupled with the use of tDCS in normal aging. Strategic memory trainings allow to improve participants' performance in the practiced task and to generalize the use of memory strategies to new materials. This Randomized Controlled Trial (RCT) aims to evaluate the effectiveness of a combined intervention associating strategic memory training with the use of tDCS. Healthy older adults and participants with subjective cognitive decline will be recruited and randomly assigned to the experimental group (strategic memory training + ACTIVE tDCS) or the control group (strategic memory training + SHAM tDCS). All participants will be evaluated on transfer and practiced tasks before (T0) and after (T1) the treatment and during follow-up visits, scheduled at 1 month (T2) and 3 months (T3) after the intervention.

DETAILED DESCRIPTION:
The use of cognitive functions such as memory is essential for the execution of daily activities and represents a crucial element for autonomy maintenance during aging. It is known that the physiological cognitive decline associated with aging also involves memory and can significantly impact the older person's independence. For these reasons, great interest has been generated by two tools that have proved to be decisive in supporting memory functions: non-invasive neurostimulation and memory training. Transcranial direct current stimulation (tDCS) is a form of noninvasive brain stimulation that modulates brain activity by employing a direct current delivered through electrodes applied to the scalp. Recently, the use of tDCS has been combined with training interventions focused on working memory in healthy older adults, providing evidence of a significant improvement in memory function when memory training is associated with the use of tDCS compared to when it is performed without it. In particular, adaptive memory trainings coupled with stimulation of the dorsolateral prefrontal cortex provide benefits that last also at follow-up visits after 1 or 3 months, especially in participants who exhibit a lower baseline performance.

While it was observed that adaptive working memory training alone is unable to modulate brain plasticity mechanisms, it was hypothesized that tDCS can modulate brain plasticity by acting through long-term potentiation (LTP) mechanisms and that it can modulate brain neurotrophic factor (BDNF), a protein that plays a relevant role in LTP.

Several adaptive memory trainings focused on working memory, which is essential for decision-making processes and daily activities.

Even if promising results have been shown so far, it appears that no study addressed the implementation of strategic memory training coupled with the use of tDCS. Adaptive trainings allow improving the performance in each task by gradually increasing its difficulty, without however resorting to teaching a strategy. Strategic memory trainings permit not only to improve participants' performance in the practiced task but also to generalize the use of memory strategies to new tasks.

Intending to prevent cognitive impairment, using these intervention methods in healthy aging and the prodromal phases can be useful. To this end, subjective cognitive decline (SCD) indeed represents an intermediate state between normal cognition and mild cognitive impairment (nMCD) and may predict the development of objective cognitive decline.

In this frame, the primary goal of this double-blind randomized controlled trial is to assess whether the application of transcranial direct current stimulation during strategic memory training (on-line neurostimulation) enhances the effect of strategic memory training. The follow-up visits allow for investigating whether eventual improvements are preserved over time and if this combined intervention affects the evolution of cognitive decline.

The treatment protocol consists of 5 sessions (2/3 session/week, 1 hour/day) of strategic memory training combined with on-line tDCS (anodic tDCS, 2mA for 20 minutes, versus sham tDCS, applied to the dorsolateral prefrontal cortex - DLPFC).

Healthy old participants will be recruited from the general population. Participants with subjective cognitive decline (SCD) are recruited from Neuropsychology/Alzheimer's Disease Assessment Unit and Neurorehabilitation Unit of IRCCS Mondino Foundation. The diagnosis of SCD is formulated based on a comprehensive neuropsychological evaluation (baseline cognitive assessment - T0) according to the guidelines presented in the literature.

At T0, the following standardized tests are used:

* Global cognitive function is assessed using Mini-Mental State Examination (MMSE);
* Cognitive reserve is assessed using Cognitive Reserve Index Questionnaire (CRIq);
* Mood is assessed using Geriatric Depression Scale (GDS).

At T0, practiced and not practiced memory tasks (Bottiroli et al., 2013) will be administered to the participants as pre-tests:

1. Associative learning;
2. List learning;
3. Name-face learning;
4. Place learning;
5. Text learning;
6. Grocery learning;

Participants who met the inclusion and exclusion criteria are enrolled and randomly assigned to the experimental group (strategic memory training + ACTIVE tDCS) or control group (strategic memory training + SHAM tDCS).

ELIGIBILITY:
Inclusion Criteria:

* MMSE ≥ 24.
* GDS < e uguale 11.
* Age between 65 and 85 years.
* Educational level ≥ 5 years.

Exclusion Criteria:

* Pre-existing cognitive impairment (e.g. aphasia, neglect).
* Dementia.
* Severe disturbances in consciousness.
* Concomitant severe psychiatric disease or other neurological conditions (e.g. depression and behavioral disorders).
* Motor or sensory diseases that may interfere with test execution or strategic memory training.

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2023-07-30 (Estimated); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Associative learning test scores | Immediately after the intervention program (T1).
  Participants are presented with 40 paired associates. Pairs consist of words chosen from Paivio, Yuille, and Madigan (1968) concreteness and imagery norms and from De Mauro, Mancini, Vedovelli, and Voghera (1993) word frequency norms. Each pair is printed in the middle of a 5 x 7 index card. The 40 cards are handed to participants, who are instructed to study the pairs for up to 20 minutes. After study, each stimulus is individually presented, and participants Are asked to write the corresponding response
Associative learning test scores | 1 month (T2) after the end of the intervention program.
  Participants are presented with 40 paired associates. Pairs consist of words chosen from Paivio, Yuille, and Madigan (1968) concreteness and imagery norms and from De Mauro, Mancini, Vedovelli, and Voghera (1993) word frequency norms. Each pair is printed in the middle of a 5 x 7 index card. The 40 cards are handed to participants, who are instructed to study the pairs for up to 20 minutes. After study, each stimulus is individually presented, and participants Are asked to write the corresponding response
Associative learning test scores | 3 months (T3) after the end of the intervention program.
  Participants are presented with 40 paired associates. Pairs consist of words chosen from Paivio, Yuille, and Madigan (1968) concreteness and imagery norms and from De Mauro, Mancini, Vedovelli, and Voghera (1993) word frequency norms. Each pair is printed in the middle of a 5 x 7 index card. The 40 cards are handed to participants, who are instructed to study the pairs for up to 20 minutes. After study, each stimulus is individually presented, and participants Are asked to write the corresponding response

SECONDARY OUTCOMES:
List learning tests scores | Immediately after the intervention program (T1).
  Participants are presented with 40 words. Words are also taken from Paivio Yuille, and Madigan (1968) and De Mauro, Mancini, Vedovelli, and Voghera (1993) norms. Each word is printed in the middle of a 5 x 7 index card. The 40 cards are handed to participants, who are instructed to study the words for up to 20 minutes. After study, participants are asked to write down as many words as they could remember (in any order) on an answer sheet.
List learning tests scores | 1 month (T2) after the end of the intervention program.
  Participants are presented with 40 words. Words are also taken from Paivio Yuille, and Madigan (1968) and De Mauro, Mancini, Vedovelli, and Voghera (1993) norms. Each word is printed in the middle of a 5 x 7 index card. The 40 cards are handed to participants, who are instructed to study the words for up to 20 minutes. After study, participants are asked to write down as many words as they could remember (in any order) on an answer sheet.
List learning tests scores | 3 months (T3) after the end of the intervention program.
  Participants are presented with 40 words. Words are also taken from Paivio Yuille, and Madigan (1968) and De Mauro, Mancini, Vedovelli, and Voghera (1993) norms. Each word is printed in the middle of a 5 x 7 index card. The 40 cards are handed to participants, who are instructed to study the words for up to 20 minutes. After study, participants are asked to write down as many words as they could remember (in any order) on an answer sheet.
Name-face learning test scores | Immediately after the intervention program (T1).
  Participants are presented with 20 black and white photographs of faces (2.75 x 4) paired with the last name printed below it. The 20 name-face cards are handed to participants, who are instructed to study the pairs for up to 20 minutes. After study, each face is individually presented, and participants are asked to write down the name that had been previously paired with it.
Name-face learning test scores | 1 month (T2) after the end of the intervention program.
  Participants are presented with 20 black and white photographs of faces (2.75 x 4) paired with the last name printed below it. The 20 name-face cards are handed to participants, who are instructed to study the pairs for up to 20 minutes. After study, each face is individually presented, and participants are asked to write down the name that had been previously paired with it.
Name-face learning test scores | 3 months (T3) after the end of the intervention program.
  Participants are presented with 20 black and white photographs of faces (2.75 x 4) paired with the last name printed below it. The 20 name-face cards are handed to participants, who are instructed to study the pairs for up to 20 minutes. After study, each face is individually presented, and participants are asked to write down the name that had been previously paired with it.
Place learning test scores | Immediately after the intervention program (T1).
  Participants are presented a map of a city. The map includes the location and name of 20 target places (e.g., bank) across the streets of an imaginary city. They are given up to 15 minutes to study, and then they have to write the position and name of places on a blank map.
Place learning test scores | 1 month (T2) after the end of the intervention program.
  Participants are presented a map of a city. The map includes the location and name of 20 target places (e.g., bank) across the streets of an imaginary city. They are given up to 15 minutes to study, and then they have to write the position and name of places on a blank map.
Place learning test scores | 3 months (T3) after the end of the intervention program.
  Participants are presented a map of a city. The map includes the location and name of 20 target places (e.g., bank) across the streets of an imaginary city. They are given up to 15 minutes to study, and then they have to write the position and name of places on a blank map.
Text learning test scores | Immediately after the intervention program (T1).
  Participants are presented with a short story with 22 major ideas (e.g., It was a quiet Sunday at Tirano railway station./ The locomotive, to which the carriages had already been coupled, was standing on the track./ The engine driver and his assistants got down to make sure everything was all right./ Some damage to the brakes...). They have up to 15 minutes to study the story, and then they are asked to recall and write down as much as possible from memory.
Text learning test scores | 1 month (T2) after the end of the intervention program.
  Participants are presented with a short story with 22 major ideas (e.g., It was a quiet Sunday at Tirano railway station./ The locomotive, to which the carriages had already been coupled, was standing on the track./ The engine driver and his assistants got down to make sure everything was all right./ Some damage to the brakes...). They have up to 15 minutes to study the story, and then they are asked to recall and write down as much as possible from memory.
Text learning test scores | 3 months (T3) after the end of the intervention program.
  Participants are presented with a short story with 22 major ideas (e.g., It was a quiet Sunday at Tirano railway station./ The locomotive, to which the carriages had already been coupled, was standing on the track./ The engine driver and his assistants got down to make sure everything was all right./ Some damage to the brakes...). They have up to 15 minutes to study the story, and then they are asked to recall and write down as much as possible from memory.
Grocery learning test scores | Immediately after the intervention program (T1).
  Participants are presented with a list of 40 grocery items (e.g., butter). Each item is printed in the middle of a 5 x 7 index card. The 40 cards are handed to participants, who are instructed to study the pairs for up to 15 minutes. In the recall phase, participants are asked to write down as many grocery items (in any order) as they could remember.
Grocery learning test scores | 1 month (T2) after the end of the intervention program.
  Participants are presented with a list of 40 grocery items (e.g., butter). Each item is printed in the middle of a 5 x 7 index card. The 40 cards are handed to participants, who are instructed to study the pairs for up to 15 minutes. In the recall phase, participants are asked to write down as many grocery items (in any order) as they could remember.
Grocery learning test scores | 3 months (T3) after the end of the intervention program.
  Participants are presented with a list of 40 grocery items (e.g., butter). Each item is printed in the middle of a 5 x 7 index card. The 40 cards are handed to participants, who are instructed to study the pairs for up to 15 minutes. In the recall phase, participants are asked to write down as many grocery items (in any order) as they could remember.

CONTACTS AND LOCATIONS:
Overall Officials: Stefano Cappa, MD, Principal Investigator — Dementia Research Center

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Antonenko D, Thams F, Grittner U, Uhrich J, Glockner F, Li SC, Floel A. Randomized trial of cognitive training and brain stimulation in non-demented older adults. Alzheimers Dement (N Y). 2022 Feb 23;8(1):e12262. doi: 10.1002/trc2.12262. eCollection 2022. PMID 35229023
- [Background] Assecondi S, Hu R, Kroeker J, Eskes G, Shapiro K. Older adults with lower working memory capacity benefit from transcranial direct current stimulation when combined with working memory training: A preliminary study. Front Aging Neurosci. 2022 Oct 10;14:1009262. doi: 10.3389/fnagi.2022.1009262. eCollection 2022. PMID 36299611
- [Background] Bottiroli S, Cavallini E, Dunlosky J, Vecchi T, Hertzog C. The importance of training strategy adaptation: a learner-oriented approach for improving older adults' memory and transfer. J Exp Psychol Appl. 2013 Sep;19(3):205-18. doi: 10.1037/a0034078. Epub 2013 Aug 26. PMID 23978160
- [Background] Grady C. The cognitive neuroscience of ageing. Nat Rev Neurosci. 2012 Jun 20;13(7):491-505. doi: 10.1038/nrn3256. PMID 22714020
- [Background] Kane MJ, Engle RW. Working-memory capacity and the control of attention: the contributions of goal neglect, response competition, and task set to Stroop interference. J Exp Psychol Gen. 2003 Mar;132(1):47-70. doi: 10.1037/0096-3445.132.1.47. PMID 12656297
- [Background] Lu H, Cheng PL, Lim BK, Khoshnevisrad N, Poo MM. Elevated BDNF after cocaine withdrawal facilitates LTP in medial prefrontal cortex by suppressing GABA inhibition. Neuron. 2010 Sep 9;67(5):821-33. doi: 10.1016/j.neuron.2010.08.012. PMID 20826313
- [Background] Park DC, Lautenschlager G, Hedden T, Davidson NS, Smith AD, Smith PK. Models of visuospatial and verbal memory across the adult life span. Psychol Aging. 2002 Jun;17(2):299-320. PMID 12061414
- [Background] Pergher V, Au J, Alizadeh Shalchy M, Santarnecchi E, Seitz A, Jaeggi SM, Battelli L. The benefits of simultaneous tDCS and working memory training on transfer outcomes: A systematic review and meta-analysis. Brain Stimul. 2022 Nov-Dec;15(6):1541-1551. doi: 10.1016/j.brs.2022.11.008. Epub 2022 Nov 29. PMID 36460294
- [Background] Reisberg B, Shulman MB. Commentary on "a roadmap for the prevention of dementia II: Leon Thal Symposium 2008." Subjective cognitive impairment as an antecedent of Alzheimer's dementia: policy import. Alzheimers Dement. 2009 Mar;5(2):154-6. doi: 10.1016/j.jalz.2009.01.011. No abstract available. PMID 19328449
- [Background] Ripp I, Emch M, Wu Q, Lizarraga A, Udale R, von Bastian CC, Koch K, Yakushev I. Adaptive working memory training does not produce transfer effects in cognition and neuroimaging. Transl Psychiatry. 2022 Dec 13;12(1):512. doi: 10.1038/s41398-022-02272-7. PMID 36513642
- [Background] Teixeira-Santos AC, Moreira CS, Pereira DR, Pinal D, Fregni F, Leite J, Carvalho S, Sampaio A. Working Memory Training Coupled With Transcranial Direct Current Stimulation in Older Adults: A Randomized Controlled Experiment. Front Aging Neurosci. 2022 Apr 12;14:827188. doi: 10.3389/fnagi.2022.827188. eCollection 2022. PMID 35493937